CLINICAL TRIAL: NCT00520338
Title: Celecoxib for Reducing Morphine Requirement After Thyroid Surgery: A Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sirilak Suksompong, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 117/2007
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Postoperative Pain; Thyroidectomy; Cyclooxygenase 2 Inhibitors
Keywords: celecoxib; postoperative pain; thyroidectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): 1. placebo
  2. celecoxib
  Interventions: Drug: celecoxib
- 1 (No Intervention): 1 placebo

INTERVENTIONS:
Drug: celecoxib — 1. placebo
  2. celecoxib 400 mg oral single dose
  Other Names: celebrex
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether celecoxib is effective in the treatment postoperative pain after thyroidectomy.

The research hypothesis:

There is a difference in postoperative morphine consumption in the first 24 hours after thyroidectomy between patients who received celecoxib or placebo.

DETAILED DESCRIPTION:
Postoperative pain has been concerned in the past few years by both the anesthesiologists ans the surgeons. COX2-inhibitors have played an important roles in postoperative pain with minimal side effects.

Comparison(s): There is a difference in postoperative morphine consumption in the first 24 hours after thyroidectomy between patients who received celecoxib and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ASA physical status I-III.
2. Scheduled for an elective thyroidectomy.
3. Body weight > or = 40kg
4. Can operate a patient-controlled analgesia (PCA) device.

Exclusion Criteria:

1. History of asthma, acute rhinitis, nasal polyps, angioneurotic edema or urticaria following the administration of aspirin or other NSAIDs.
2. Known hypersensitivity to morphine or sulfonamides.
3. History of hepatic dysfunction.
4. Creatinine clearance < 30ml/min.
5. History of bleeding tendency.
6. History of gastrointestinal bleeding or active peptic ulcer.
7. Known case of inflammatory bowel disease.
8. Patient with severe heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The patients' total amount of morphine requirement in the first 24 hour. | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Department of anesthesiology. Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand